CLINICAL TRIAL: NCT03747185
Title: Corticospinal Excitability of Deep Back and Abdominal Muscles in Individuals With History of Clinical Lumbar Instability
Brief Title: Corticospinal Excitability of Deep Back and Abdominal Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Peemongkon Wattananon, Principal investigator, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/128.2906
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Instability; Back; Tightness of Back Muscles
Keywords: Clinical lumbar instability; History of low back pain; Corticospinal excitability; Stretching exercise; Movement system impairment

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either stretching exercise with lumbopelvic stiffening technique or lumbopelvic relaxing technique. They will be provided a 2-day wash-out period. Then, participants will cross-over to another technique.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor and investigator will be blinded to the random order. This process will be handled by the research manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbopelvic stiffening technique (Experimental): Hamstring muscle stretching with lumbopelvic stiffening technique.
  Interventions: Other: Lumbopelvic stiffening technique; Other: Lumbopelvic relaxing technique
- Lumbopelvic relaxing technique (Active Comparator): Hamstrings muscle stretching with lumbopelvic relaxing technique.
  Interventions: Other: Lumbopelvic stiffening technique; Other: Lumbopelvic relaxing technique

INTERVENTIONS:
Other: Lumbopelvic stiffening technique — Participants will stretch the hamstrings muscle in standing position with lumbopelvic stiffening technique. Fifteen percent of the body weight will be used to standardize stretching force. During stretching protocol, the participants will be instructed to face the hydraulic table with the hips square, maintain trunk straight up and look straight ahead. Researcher commands "during adjusting the bed up, please tense the back rigid". After that, hydraulic bed will be lifted up until force reaches 15 percent of the body weight. Participant will perform 30 seconds/repetition for 4 repetitions with 15 seconds rest between repetitions.
Other: Lumbopelvic relaxing technique — Participants will be instructed to face the hydraulic table with the hips square, maintain trunk straight up and look straight ahead. The researcher commands "During adjusting the bed up, please relax the back". The hydraulic bed will be lifted up until force reaches 15 percent of the body weight. Participant will perform 30 seconds/repetition for 4 repetitions with 15 seconds rest between repetitions.

SUMMARY:
This study aims to understand the roles of corticospinal excitability in controlling the trunk movement, and the clinical utility of clinical observation, as well as the effect of lumbopelvic stabilization during hamstrings muscle stretching.

DETAILED DESCRIPTION:
This study will use a sample of convenience between the ages of 20 and 40. Subjects with and without history of low back pain will be recruited by flyers posted in university physical therapy clinics in 2 locations, as well as word of mouth from subjects and friends. Subjects who are interested in participation will undergo a screening process using inclusion-exclusion criteria checklist and receive brief information regarding the study. If the participants meet all inclusion criteria, the consent process will be performed. To ensure the participants understand the study, the participants will be simply asked regarding the study (i.e. objectives, benefits, etc.) before signing the consent form. Total data collection including intervention between pre- and post-intervention will take approximately 2 hours.

After obtaining the written informed consent, all participants will fill out the information sheet for demographic data. Participant will have the right to refuse answering the demographic questionnaire, but the participants can participate in biomechanical data collection. Then, participants will asked to remove the metal accessories that could influence the electromagnetic field, change the cloth to lab tank top and shorts to expose the lower back and right knee, and wear the shoes throughout the test protocol. The body landmarks will be identified. These landmarks include 1) lumbar spine level 1 (L1), 2) sacrum level 2 (S2), 3) lateral epicondyle of right (RE) and left (LE) knees, and 4) head of fibula of right (RF) and left (LF) leg. These locations will be used to place motion sensors for outcome measures. The preparation process will take approximately 10 minutes.

The subjects will stand in a natural stance with arms down by sides. The participants will be instructed to perform functional movements including active forward bend, right and left straight leg raise tests, right and left hip abduction with knee flexion tests, quadruped backward rock test, prone with right and left knee flexion tests, prone with right and left hip internal/external rotation tests, prone with right and left hip extension tests. Each subject performs 2 trials of 3 consecutive repetitions of each functional movement tests. Heart rate and rating of perceive exertion (RPE) will be monitored after each functional movement tests. Two physical therapists (PT-A and PT-B), who are blinded to the group membership, will simultaneously observe and independently rate aberrant movement patterns. After physical therapists completing the clinical observation, the participants will hand the rating form to the principal investigator to input into a spreadsheet for further analysis. These data will be used to determine inter-rater reliability and diagnostic accuracy of clinical observation of aberrant movement patterns during functional movements to identify individuals with a history of CLI. The clinical observation will take about 20 minutes.

Prior to performing SLR, motion sensors will be placed on the subject's body landmarks. Subjects will be asked to perform one repetition of active forward bend, while motion data are simultaneously collected. Then, subjects will be asked to lay on the treatment table in supine position. PT-A will perform passive SLR, and maximal angle will be recorded. This SLR test is intended to determine whether the subject has a sign of CLI, rather than to assess neural tension (to rule out HNP and dural tension) or hamstrings muscle length. In participants with clinical lumbar instability, pelvis/hip will not be stabilized when performing passive SLR. In this case, when pelvis/hip has reached its restriction by hamstrings muscle tightness, lumbar spine would easily allow compensatory motion. Thus, leg raising greater than 91° would indicate clinical lumbar instability. This test is differed from hamstrings muscle tightness (passive knee extension in supine with 90° hip flexion position). This test the clinician will fix the pelvic/hip at 90°; therefore, compensatory motion from pelvis/hip will be minimized. After that, PT-A will perform hamstrings muscle length test. Subjects will be first asked to lay on the treatment table with tested hip and knee in 90 degrees flexion. PT-A will passively extend subject's knee to maximal tolerable point. Angle in sagittal plane between lateral epicondyle and head of fibula sensors will be measured to represent hamstrings muscle length. PT-A will perform additional clinical examination including modified Thomas test (muscle length test for iliopsoas, quadriceps, hip abductor, and hip adductor muscles), Ober's test (muscle length test for tensor fascia latae muscle), as well as abdominal and back muscle strength test assessed by a handheld dynamometer. These outcome measures will be assessed for baseline. To reduce the risk of muscle fatigue, the investigators will monitor heart rate and verbally ask the RPE during the test, and provide adequate resting period between repetitions. The clinical examination will take approximately 10 minutes.

After clinical data collection, the subjects will undergo corticospinal excitability measurement using transcranial magnetic stimulation (TMS). The investigator will identify transversus abdominis muscle (2 cm medial and 2 cm inferior to anterior superior iliac spine on the inguinal line), and lumbar multifidus muscle (2 cm lateral to lumbar spinous process of level 4). These locations will be used for EMG electrode placement. Before placing surface EMG electrodes, the skin will be lightly abraded using abrasive paper and cleaned using cotton with alcohol to lower the skin impedance. Electrodes will be aligned parallel to the muscle fibers. Then, Subjects will be seated comfortably in a reclined chair with both arms supported. The participants will be asked to wear a swim cap used to identify stimulation areas for transverse abdominis and lumbar multifidus muscles. The investigator will use a double cone coil to find the hotspot for both ipsilateral and contralateral to the pain in each muscle. Figure 1 illustrates TMS set up. After corticospinal excitability measurement, subjects will be randomly assigned into 2 groups (lumbopelvic stabilization, LPS and lumbopelvic relaxation, LPR). The TMS data collection will take approximately 60 minutes.

The subjects in both groups will perform hamstrings muscle stretching in standing position. The participants will be asked to place the heel on the tested leg on the compression load cell mounted on the adjustable treatment table. The adjustable treatment table will be initially set at the subject's knee level. Treatment table will gradually move up until force at the heel reaches 15% of the body weight. This standardized force will be controlled by the compression load cell. Our preliminary study indicates that 15% of the body weight is the maximal stretching force in which subjects have reported very hard level of exertion (16-18 out of 20) on RPE during stretching exercise. During applying stretching force, subjects in LPS will be asked to keep the lumbar and pelvic positions as rigid as possible without holding the breath, while subjects in LPR will be asked to relax the lumbopelvic region and do not hold against stretching force. Each subject will perform 4 repetitions of 30-second stretching with 15 seconds rest between repetitions.

After the intervention, the subjects will be reassessed for lumbopelvic motion during forward bend and hamstrings muscle length test. The intervention and reassessment process will take approximately 20 minutes. The data at baseline and post-intervention will be used to determine the effect of lumbopelvic stabilization during hamstring muscle stretching in individuals with and without a history of CLI. In addition, the investigator will call each subject for 1-year follow up to check whether subjects have any episode of low back pain and how often the participants have low back pain.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for individuals without a history of clinical lumbar instability.

  1. Between the ages of 20 and 40
  2. No history of LBP that interferes with activities of daily living and/or required treatment
* The inclusion criteria for individuals with a history of clinical lumbar instability.

  1. Between the ages of 20 and 40
  2. A recurrent pattern of LBP at least two episodes that interfered with activities of daily living and/or required treatment
  3. Presenting aberrant movement pattern during active forward bend test
  4. Passive straight leg raising test (SLR) greater than 91 degrees
  5. Having hamstrings muscle tightness of both legs (passive knee extension in supine with 90° hip flexion position greater than 20 degrees)

Exclusion Criteria:

1. History of seizure for either the subject or any family member
2. Implanted pacemaker
3. Clinical signs of systemic disease
4. Definitive neurologic signs including pain, weakness or numbness in the lower extremity
5. Previous spinal surgery
6. Diagnosed osteoporosis, severe spinal stenosis, and/or inflammatory joint disease
7. Any lower extremity condition that would potentially alter trunk movement
8. Vestibular dysfunction
9. Extreme psychosocial involvement
10. Body mass index (BMI) greater than 30 kg/m2
11. Active treatment of another medical illness that would preclude participation in any aspect of the study
12. Menstruation or pregnancy (for female subject)
13. Diagnosed herniated nucleus pulposus (HNP)
14. Pain medication usage (e.g., NSAID)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Resting and active motor threshold | These data will be collected at baseline only.
  Resting and active motor threshold (MT) for ipsilateral and contralateral responses for transverse abdominis and lumbar multifidus muscles.
Motor evoke potentials | These data will be collected at baseline only.
  Motor evoke potentials (MEP) for transverse abdominis and lumbar multifidus muscles.
Center of gravity of Topography | These data will be collected at baseline only.
  Center of gravity coordinate of Topography of transverse abdominis and lumbar multifidus muscles.
Volume of Topography | These data will be collected at baseline only.
  Volume of Topography of transverse abdominis and lumbar multifidus muscles.
Clinical observation of aberrant movement. | These data will be collected at baseline only.
  Clinical observation of aberrant movement patterns during functional movement will be performed by two physical therapists.
Motion data. | These data will be measure at baseline and immediately after receiving stretching exercise technique.
  Clinical motion analysis system will be used to measure lumbar, pelvic, lumbopelvic, and knee motions. This system is composed of triple axis accelerometers (MPU6050, China), data acquisition board (Arduino Uno R3, Italy), and a LabVIEW software version 2012 (National Instrument, USA). The system will be used to measure pre- and post-intervention of angle of lumbar, pelvic, and lumbopelvic motions through a custom LabVIEW program at 100 Hz.

SECONDARY OUTCOMES:
Passive straight leg raising to test clinical lumbar instability | These data will be collected at baseline only.
  Clinical tests will be performed at the baseline because they could be a potential confounding factor.
Muscle length based on modified Thomas and Trendelenburg test | These data will be collected at baseline only.
  Clinical tests will be performed at the baseline because they could be a potential confounding factor.
Abdominal and back muscle strength . | These data will be collected at baseline only.
  Clinical tests will be performed at the baseline because they could be a potential confounding factor.
1-year follow-up. | 1 year after data collection.
  Participants will be call to check whether they have any episode of low back pain and how often they have low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, PhD, Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The IPD of this study will be shared upon official request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The supporting information will be sent upon official request.
Access Criteria: Having an official written request.

REFERENCES:
- [Background] Tsao H, Galea MP, Hodges PW. Reorganization of the motor cortex is associated with postural control deficits in recurrent low back pain. Brain. 2008 Aug;131(Pt 8):2161-71. doi: 10.1093/brain/awn154. Epub 2008 Jul 18. PMID 18669505
- [Background] Tsao H, Tucker KJ, Hodges PW. Changes in excitability of corticomotor inputs to the trunk muscles during experimentally-induced acute low back pain. Neuroscience. 2011 May 5;181:127-33. doi: 10.1016/j.neuroscience.2011.02.033. Epub 2011 Feb 17. PMID 21333720
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] Sahrmann S, Azevedo DC, Dillen LV. Diagnosis and treatment of movement system impairment syndromes. Braz J Phys Ther. 2017 Nov-Dec;21(6):391-399. doi: 10.1016/j.bjpt.2017.08.001. Epub 2017 Sep 27. PMID 29097026
- [Background] Jandre Reis FJ, Macedo AR. Influence of Hamstring Tightness in Pelvic, Lumbar and Trunk Range of Motion in Low Back Pain and Asymptomatic Volunteers during Forward Bending. Asian Spine J. 2015 Aug;9(4):535-40. doi: 10.4184/asj.2015.9.4.535. Epub 2015 Jul 28. PMID 26240711